CLINICAL TRIAL: NCT02372084
Title: A Phase I, Open-label, Multi-center, Single Dose, Parallel Group Study to Evaluate the Pharmacokinetics and Safety of Osilodrostat (LCI699) in Subjects With Impaired Hepatic Function Compared to Subjects With Normal Hepatic Function
Brief Title: A Phase 1 Study of Osilodrostat (LCI699) in Healthy Volunteers and Subjects With Impaired Hepatic Function
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CLCI699C2103
Record Dates: First submitted 2015-02-23; First posted 2015-02-26 (Estimated); Last update posted 2020-12-19 (Actual); Status verified 2020-05

CONDITIONS: Hepatic Impairment
Keywords: Hepatic impairment,; osilodrostat,; LCI699
MeSH Terms: interventions — Osilodrostat

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- osilodrostat (LCI699) (Experimental): Each participant will undergo a 28-day screening/baseline period (day -28 to day -1), followed by a 5 day treatment period (a single 30 mg dose of LCI699 ( Day 1) with 5 days of PK sample collection).
  Interventions: Drug: osilodrostat

INTERVENTIONS:
Drug: osilodrostat
  Other Names: LCI699

SUMMARY:
To assess the pharmacokinetics of a single oral dose of osilodrostat (LCI699) 30 mg in subjects with mild, moderate and severe hepatic impairment compared with subjects with normal hepatic function.

ELIGIBILITY:
Inclusion Criteria:

* Weight ≥50 kg and BMI between 18-38kg/m2.
* Stable liver cirrhosis and evidence of hepatic impairment.
* Free of significant medical disorders unrelated to underlying hepatic impairment

Exclusion Criteria:

* History of any surgical or medical condition which might significantly alter the absorption, distribution, metabolism or excretion of drugs
* Subjects with ongoing alcohol or drug abuse
* Symptoms or history of encephalopathy (Grade 2 or above)
* History or presence of liver disease or liver injury (healthy volunteers only)
* History or presence of impaired renal function
* Clinical evidence of severe ascites.
* Total Bilirubin > 6 mg/dL,
* Subjects with a serum free cortisol test results that is below the lower limit of normal (based on central laboratory) during the screening period
* Concomitant use of a drug that is a strong inducer of the CYP3A4/5 pathway

Other protocol-defined inclusion/exclusion criteria may apply -

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 33 (Actual)
Dates: Start 2015-04-21 (Actual); Primary Completion 2016-05-19 (Actual); Study Completion 2016-05-19 (Actual)

PRIMARY OUTCOMES:
Pharmacokinetics (PK) of a single dose of 30 mg osilodrostat: AUClast | Predose (Day 0) , and at timepoints 0.5, 1, 1.5, 2, 3,4, 6, 8, 12, 24, 36, 48, 72, 96 hours post dose.
  To assess the influence of hepatic impairment on the pharmacokinetics (PK) of LCI699i in subjects with varying degrees of hepatic impairment compared to subjects with normal hepatic function.
PK of a single dose of 30 mg osilodrostat: AUCinf | Predose (Day 0) , and at imepoints 0.5, 1, 1.5, 2, 3,4, 6, 8, 12, 24, 36, 48, 72, 96 hours post dose.
  To assess the influence of hepatic impairment on the pharmacokinetics (PK) of LCI699i in subjects with varying degrees of hepatic impairment compared to subjects with normal hepatic function.
PK of a single dose of 30 mg osilodrostat: Cmax | Predose (Day 0) , and at timepoints 0.5, 1, 1.5, 2, 3,4, 6, 8, 12, 24, 36, 48, 72, 96 hours post dose.
  To assess the influence of hepatic impairment on the pharmacokinetics (PK) of LCI699i in subjects with varying degrees of hepatic impairment compared to subjects with normal hepatic function.
PK of a single dose of 30 mg osilodrostat: T1/2 | Predose (Day 0) , and at timepoints 0.5, 1, 1.5, 2, 3,4, 6, 8, 12, 24, 36, 48, 72, 96 hours post dose.
  To assess the influence of hepatic impairment on the pharmacokinetics (PK) of LCI699i in subjects with varying degrees of hepatic impairment compared to subjects with normal hepatic function.
PK of a single dose of 30 mg osilodrostat: CL/F | Predose (Day 0) , and at timepoints 0.5, 1, 1.5, 2, 3,4, 6, 8, 12, 24, 36, 48, 72, 96 hours post dose.
  To assess the influence of hepatic impairment on the pharmacokinetics (PK) of LCI699i in subjects with varying degrees of hepatic impairment compared to subjects with normal hepatic function.
PK of a single dose of 30 mg osilodrostat: Vz/F | Predose (Day 0) , and timepoints 0.5, 1, 1.5, 2, 3,4, 6, 8, 12, 24, 36, 48, 72, 96 hours post dose.
  To assess the influence of hepatic impairment on the pharmacokinetics (PK) of LCI699i in subjects with varying degrees of hepatic impairment compared to subjects with normal hepatic function.

SECONDARY OUTCOMES:
The relationship between PK parameters (Cmax and AUC) and baseline hepatic function parameters namely; total bilirubin, albumin, INR (or prothrombin, if INR unavailable) | Predose ( Day 0) and at timepoints 0.5, 1, 1.5, 2, 3,4, 6, 8, 12, 24, 36, 48, 72, 96 hours post dose.
  To evaluate the relationship between hepatic function parameters and pharmacokinetics.
Number of participants with adverse events (AEs) | Pre-treatment, during treatment (Day 1) and 30 days post treatment.
  This will be assessed using laboratory abnormalities, ECG and vital sign assessments of a single 30 mg dose of LCI699

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (3):
- United States (3):
  - University of Miami / Clinical Research Services, Inc. Boynton Beach, Miami, Florida
  - Orlando Clinical Research Center, Orlando, Florida
  - DaVita Clinical Research, Minneapolis, Minnesota

REFERENCES:
- See also: Novartis results database — https://www.novctrd.com/ctrdweb/trialresult/trialresults/pdf?trialResultId=16087